CLINICAL TRIAL: NCT04107337
Title: Randomized Study of the Effect of Vocal Exercises With Straw on Aerodynamic Parameters of Voice (Pressure, Flow) in Dysodic Singers With Nodules
Brief Title: Effect of Vocal Exercises With Straw on Aerodynamic Parameters of Voice (Pressure, Flow) in Dysodic Singers With Nodules
Acronym: DYSODIE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL19_0262
Record Dates: First submitted 2019-08-01; First posted 2019-09-27 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-09

CONDITIONS: Dysodia; Vocal Disorders
Keywords: Dysodia; Singers; Straw; Estimated subglottal pressure; Aerodynamic measurements; Oral airflow
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Intervention Model Description: 1. Experimental group (N=10): vocal work session based on semi-occluded vocal-tract exercises with a straw.
  2. Control group (N=10): the second group acting as control group will perform a vocal work session based on open mouth exercices (vocalizations).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group (N=10): this group will conduct a vocal work session based on semi-occluded vocal-tract exercises with a straw.
  Interventions: Other: Vocal work session with straw exercises
- Control group (Other): Control group (N=10): the second group acting as control group will perform a vocal work session based on open mouth exercices (vocalizations).
  Interventions: Other: Vocal work session with open mouth exercises

INTERVENTIONS:
Other: Vocal work session with straw exercises — * Voice assessment: A questionnaire on the subject's voice biography will be sent to the subject at the moment of inclusion.
  * Vocal exercises during 10 minutes : (1 minute) Checking the posture ; (1 minute) Control of the management of breath in the straw ; (1 minute) Phonation in the straw ; (2 minutes) Make a siren in the straw ; (4 minutes) Vocalizations in the straw on the arpeggio of Rossini.
  This working session will be preceded and followed by the same 10-minutes voice assessment focusing on aerodynamic parameters.
  Arms: Experimental group
Other: Vocal work session with open mouth exercises — * Voice assessment: A questionnaire on the subject's voice biography will be sent to the subject at the moment of inclusion.
  * Vocal exercises during 10 minutes : (1 minute) Checking the posture ; (1 minute) Control of the management of breath on a [f] with open mouth ; (1 minute) Phonation on the vowel [a] with open mouth ; (2 minutes) Make a siren on the vowel [a] with open mouth ; (4 minutes) Vocalizations on the vowel [a] on the arpeggio of Rossini with open mouth.
  This working session will be preceded and followed by the same 10-minutes voice assessment focusing on aerodynamic parameters.
  Arms: Control group

SUMMARY:
Singers are over-represented in phoniatric consultations; they present increased risk of developing voice disorders. The most common lesion found in singers is nodule. It comes from vocal straining characterized by the use of a pressed phonation mode, resulting in an increase subglottal pressure and a decrease flow rate. Voice therapy aims to restore a more relaxed phonation. There is a growing interest in semi-occluded vocal tract exercises with a straw in therapy; they have positive effects, particularly in terms of aerodynamic parameters such as subglottal pressure and oral airflow. After these exercises, subglottal pressure decreases and oral airflow increases. In other words, patient adopts a more relaxed phonation mode. Several studies have investigated the effect of these straw exercises on dysphonic patients i.e. on speaking voice; no study to date has explored the effect of these exercises on dysodic subjects i.e. on singing voice.

The aim of this study is to evaluate the impact of straw exercises compared to open-mouth exercises on aerodynamic parameters in dysodic women singers with nodules.

DETAILED DESCRIPTION:
Singers are over-represented in phoniatric consultations; they present increased risk of developing voice disorders whether they are amateurs or professionals. They represent a specific population among phoniatric patients because of their increased sensitivity to the slightest vocal change that makes them consult earlier than non-singers. In addition, their complaints are specific to singing voice.

In phoniatrics, at the CHU Gui de Chauliac in Montpellier, singers (amateurs and professionals) represent one third of phoniatric patients. 80% of them are diagnosed with dysodia. Dysodia refers to singing voice disorders, in the same way as dysphonia refers to speaking voice disorders.

Dysodia results in a variety of symptoms. Acoustic signs are the most numerous: tonal anomalies (lack of accuracy, reduction of vocal range); dynamic anomalies (problem to sing softly or loudly); timbre abnormalities (vibrato problems, strained voice , roughness, difficulties on attacks). Dysodia also results in respiratory disorders, physical signs, psychological consequences and damage to hedonistic properties (loss of comfort, vocal endurance, musicality).

It can reach amateur or professional singers. For professional singers, voice is the main working tool. When they have dysodia, professional difficulties can be temporary or even lead to the loss of work. In addition, dysodia can lead to financial loss and well-documented anxiety. For amateur singers, dysodia hinders their musical practice, thus limiting the recognized benefits of choral singing on cohesion, social integration and personal development.

Prevalence of dysodia is higher among women. This vocal disorder is most often associated with laryngeal pathology. Nodular lesions are most common in singers as in general population. Nodules are the consequence of vocal straining, also known as vocal hyperfunction.

Singing means learning, more or less finely, depending on the level of training and singing style, coordination between breath, vocal fold vibrations and resonators, the so-called pneumo-phono-resonant adaptations. To have balanced phonation, singer must properly dose the air pressure he applies under his vocal folds, have a sufficient flow rate and adapt muscular tension of the vocal folds (neither too strain nor too loose). In this mode of phonation, voice resonates without difficulty. On the other hand, during vocal straining, singer will put too much subglottal pressure decreasing flow rate, which creates a laryngeal tightening and can eventually cause nodules. The pressure threshold required to initiate a sound (phonation pressure threshold) is then increased. Vocal gesture is therefore inappropriate and the voice becomes ineffective.

After diagnosis of dysodia and vocal assessment to identify the patient's difficulties, the patient is referred to speech-language pathologist for voice therapy. According to the vocal difficulties identified, speech therapist defines the therapeutic objectives that will be adapted to each patient and individualized according to the diagnosis, the singer's profile, but also his objectives and his investment. Voice therapy aims not only to prevent the onset or aggravation of vocal disturbances but also to remove or compensate for voice limitations by reconditioning vocal gesture to make it more effective. In the case of nodular lesions, voice therapy therefore aims to reduce vocal straining.

There is no specific therapeutic tool for singers. As in speaking voice, speech-language pathologist uses technical aids as well as indirect and direct therapies. The main technical aid proposed is amplification of voice with a microphone in the event of vocal misuse or abuse, i.e. when the vocal load is too high. Indirect therapy consists of giving vocal hygiene advice, in order to eliminate causes of voice disorder and to establish a vocal economy program with the patient. On the other hand, direct therapy consists in directly modifying vocal gesture through vocal exercises. This therapy is based on the premise that the subject has acquired an inappropriate vocal gesture that the therapist identifies and corrects through vocal exercices. Direct therapy is based on three successive steps: i) rehabilitation of respiratory gesture, ii) work on a vocal emission without associated tension, so as to eventually reduce laryngeal lesions, and iii) awareness of the role of resonance cavities.

Concerning work of vocal emission, to reduce vocal straining, many therapies are based on semi-occluded vocal tract exercises, also called physiological exercises. They include labial and lingual trills (lip and tongue vibration), nasal consonants, voiced fricative consonants, kazoo as well as tubes or straws. Straw exercises are the most reproducible due to the precise calibration of occlusion. Montpellier University Hospital is the national leader in the development of these straw exercises in France, with a particular focus on flow control during the exercises.

The purpose of these exercises is to teach the patient to use proper air pressure and flow while singing. Several studies are investigating effects of these straw exercises on aerodynamic parameters of subglottal pressure, phonation pressure threshold and oral airflow. It appears that:

* straw exercises reduce estimated subglottal pressure. For non-singers, this is true after 15 minutes of exercises as well as after 8 rehabilitation sessions. For singers, results are more variable and concern only singers without voice disorders. No studies have explored effect of straw exercises on estimated subglottal pressure in dysodic singers.
* straw exercises lower phonation threshold pressure (PTP). Most studies find a decrease in PTP after straw exercises, either in non-singer patients with speaking voice disorders or in choristers without voice disorders. No studies have explored effect of straw exercises on PTP in dysodic singers.
* Literature does not provide information on impact of straw exercises on oral airflow. In euphonic subjects (without vocal disorder), whether singers or not, majority of studies find an increase in airflow after straw exercises. Only one study found no difference in airflow after straw exercises, while airflow increased after vocal exercises without straw (vocalized). In dysphonic patients, no difference in flow rate is observed after straw exercises. No studies have explored effect of straw exercises on airflow in dysodic singers.

Thus, no study to date has explored effect of straw exercises on aerodynamic parameters (estimated subglottal pressure, PTP, oral airflow) in dysodic singers. Singers are often targeted as a study population because of their familiarity with semi-occluded exercises but not to further explore singing voice. For example, in a study only one frequency is tested (pitch and comfortable intensity), so singing voice is not further explored. However, the economic and psychological impact of dysodia, particularly among professionals, is well described in the literature.

In this project the investigator want to fill this gap by studying the singing voice effect of straw exercises on the estimated subglottal pressure, PTP and oral airflow in dysodic women singers. Do straw vocal exercises modify aerodynamic behaviour of dysodic women singers with nodules after a rehabilitation session? Based on results of literature for speaking and singing non-pathological voice, the investigator hypothesize that the estimated subglottal pressure and PTP will decrease after straw exercise session while they will remain constant after open mouth exercise session. Meanwhile, the investigator hypothesize that oral airflow will increase following straw exercises while it will remain constant after open-mouth exercises.

ELIGIBILITY:
Inclusion Criteria:

* be a singer
* being female
* be over 18
* have a diagnosis of dysodia associated with vocal compelling behavior. This diagnosis is made by the investigative phoniatrist coordinator of the study during the phoniatric consultation.
* have signed the written informed consent.
* be affiliated or beneficiary of a social security scheme.

Exclusion Criteria:

* have hearing problems
* Persons deprived of their liberty, protected adults or vulnerable persons
* Pregnant and / or lactating woman

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-25 (Estimated); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
Aerodynamic data : estimated subglottal pressure | before vocal exercices
  Estimated subglottal pressure (values in hPa)
Aerodynamic data : estimated subglottal pressure | after vocal exercices
  Estimated subglottal pressure (values in hPa)

SECONDARY OUTCOMES:
Aerodynamic data : phonation pressure threshold | before vocal exercices
  Phonation pressure threshold (values in hPa)
Aerodynamic data : phonation pressure threshold | after vocal exercices
  Phonation pressure threshold (values in hPa)
Aerodynamic data : oral airflow rate | before vocal exercices
  oral airflow rate (values in l/s)
Aerodynamic data : oral airflow rate | after vocal exercices
  oral airflow rate (values in l/s)

CONTACTS AND LOCATIONS:
Locations (1):
- Gui de Chauliac Hospital, Montpellier, Herault, France